CLINICAL TRIAL: NCT05836025
Title: Effect of Rapamycin in Ovarian Aging
Acronym: Rapamycin
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Samuel Zev Williams, Associate Professor of Obstetrics and Gynecology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAU1074
Record Dates: First submitted 2023-04-17; First posted 2023-05-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Perimenopausal
Keywords: Premenopausal; Perimenopause; Fertility; Women's health
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rapamycin (Experimental): Participants randomized to the treatment arm will receive 5mg/week of rapamycin orally, for 12 weeks (3 months).
  Interventions: Drug: Rapamycin
- Placebo (Placebo Comparator): Participants randomized to the placebo arm will receive placebo orally, for 12 weeks (3 months).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rapamycin — 5mg/week of rapamycin orally for 12 weeks
  Arms: Rapamycin
Other: Placebo — 5mg/week of placebo orally for 12 weeks
  Arms: Placebo

SUMMARY:
The investigators are proposing a prospective, randomized, double-blind, placebo-controlled pilot study assessing the ability of low-dose rapamycin to delay ovarian aging in women. Animal studies have shown the potential of rapamycin in slowing or reversing some age-associated pathways.

DETAILED DESCRIPTION:
One of the earliest and most profound changes associated with human aging is the rapid decline in ovarian follicular activity and reproductive capacity. Beginning around age 35, fertility rates decline as the number and quality of oocytes fall, culminating in the onset of menopause around age 51. The onset of menopause has profound socioeconomic, quality of life, and health implications, including increasing the risks of cardiovascular disease, osteoporosis, cognitive decline and dementia. While human lifespan has increased, the age of menopause has remained largely unchanged, leaving more women living an ever-larger proportion of their lives in a postmenopausal state. The narrow reproductive window adds socioeconomic pressure on women to complete childbearing within a limited timeframe, or preserve their fertility with egg or embryo freezing. The investigators and others have demonstrated that rapamycin can delay ovarian aging in mice.

The purpose of this pilot study is to determine whether the same may be true in humans. Extending the reproductive lifespan will reduce the time pressure on women to complete childbearing and will allow more women to spend more of their lives in the premenopausal status and delay the negative healthy consequences of menopause.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 35-45 years
* In the menopausal transition stage -3a
* Have been unable to conceive based on diminished ovarian reserve and who have failed to develop any euploid embryos with IVF or who do not desire to conceive within the next 1.5 years
* Have regular menstrual periods (with less than 7 days of variability)
* Early follicular phase follicle stimulating hormone (FSH) levels ] < 20 mIU/mL
* Anti-müllerian hormone (AMH) levels of >0.1 ng/mL
* Antral Follicle Counts (AFC) of >3

Exclusion Criteria:

* Women with irregular menstrual cycles
* Severe ovarian deficiency, or with no evidence of remaining follicles
* Kidney or liver disease
* Any significant medical disease, including cancer
* Contraindications to receiving rapamycin

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Measure of Ovarian Reserve | Up to 1 year
  Ovarian reserve will be determined using AMH

SECONDARY OUTCOMES:
TVU | Up to 1 year
  TVUs will be used to measure follicle growth
Estradiol (E2) Level | Day 21 of menstrual cycle
  Estradiol levels will be measured.
FSH Level | Day 21 of menstrual cycle
  Follicle stimulating hormone (FSH) levels will be measured.
Klotho Level | Day 21 of menstrual cycle
  Klotho levels will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z. Williams, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States